CLINICAL TRIAL: NCT03822351
Title: A Phase 2 Open-label, Multicenter, Randomized, Multidrug Platform Study of Durvalumab (MEDI4736) Alone or in Combination With Novel Agents in Subjects With Locally Advanced, Unresectable (Stage III) Non-small Cell Lung Cancer (COAST)
Brief Title: Durvalumab Alone or in Combination With Novel Agents in Subjects With NSCLC
Acronym: COAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9108C00001; 2018-002931-35 (EudraCT Number)
Record Dates: First submitted 2018-12-10; First posted 2019-01-30 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Stage III Non-small Cell Lung Cancer; Unresectable
Keywords: Locally Advanced NSCLC; Non-small Cell Lung Cancer; Cancer; Lung; Unresectable; Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — durvalumab; monalizumab

STUDY DESIGN:
Intervention Model Description: At study onset subjects will be randomized equally to all study treatment arms open for enrollment and will remain on study treatment for up to 12 months.
  Study treatment will be discontinued upon disease progression, unacceptable toxicity, or other reason. The treatment arms are Control Arm, Arm A and Arm B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control Arm (Durvalumab monotherapy) (Experimental): durvalumab IV
  Interventions: Drug: Durvalumab
- Arm A (durvalumab + oleclumab): (Experimental): durvalumab IV and oleclumab IV
  Interventions: Drug: Durvalumab + Oleclumab
- Arm B (durvalumab + monalizumab) (Experimental): durvalumab IV and monalizumab IV
  Interventions: Drug: Durvalumab + Monalizumab

INTERVENTIONS:
Drug: Durvalumab + Oleclumab — Durvalumab + Oleclumab
  Other Names: Durvalumab (MEDI-4736); Oleclumab (MEDI-9447)
  Arms: Arm A (durvalumab + oleclumab):
Drug: Durvalumab — Durvalumab
  Other Names: Durvalumab (MEDI-4736)
  Arms: Control Arm (Durvalumab monotherapy)
Drug: Durvalumab + Monalizumab — Durvalumab + Monalizumab
  Other Names: Durvalumab (MEDI-4736); Monalizumab (IPH2201)
  Arms: Arm B (durvalumab + monalizumab)

SUMMARY:
The purpose of this study is to compare the clinical activity of durvalumab alone vs durvalumab in combination with novel agents. The overall study goal is early identification of novel durvalumab combinations that are more active than durvalumab alone in the treatment of patients with unresectable, Stage III NSCLC who have not progressed after cCRT.

DETAILED DESCRIPTION:
Study D9108C00001 (COAST) is a Phase 2, open-label, multicenter, randomized multidrug platform study assessing the efficacy and safety of durvalumab alone vs durvalumab in combination with novel agents in subjects with locally advanced, unresectable, Stage III non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Main Inclusion Criteria:

1. Written informed consent and any locally required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluation
2. Age 18 years or older
3. Body weight ≥ 35 kg
4. Subjects must have histologically or cytologically documented NSCLC who present with locally advanced, unresectable, Stage III disease
5. Subjects must have completed, without progressing, definitive cCRT within 42 days prior to being randomized into the study
6. Provision of tumor tissue sample, when available, from original diagnosis obtained before initiation of chemoradiotherapy
7. Life expectancy ≥ 12 weeks
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
9. Subjects must have at least one previously irradiated tumor lesion that can be measured by RECIST v1.1

Main Exclusion Criteria:

1. Mixed small cell and non-small cell lung cancer histology
2. Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug
3. Prior exposure to any anti-PD1, anti-PD-L1, or anti-CTLA4 antibody for treatment of NSCLC
4. Subjects with history of ≥ Grade 2 pneumonitis from prior chemoradiation therapy
5. Subjects with a history of venous thrombosis within the past 3 months
6. Subjects with history of myocardial infarction, transient ischemic attack, or stroke in the past 6 months
7. Congestive heart failure
8. Active or prior documented autoimmune or inflammatory disorders
9. History of active primary immunodeficiency
10. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
11. History of allogenic organ transplantation
12. QTcF interval ≥ 470 ms
13. History of another primary malignancy
14. Concurrent enrollment in another clinical study [concurrent enrollment in an observational (non-interventional) clinical study or during the follow-up period of an interventional study is permitted]
15. Females who are pregnant, lactating, or intend to become pregnant during their participation in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (27):
  - Research Site, Anaheim, California
  - Research Site, Duarte, California
  - Research Site, Sacramento, California
  - Research Site, New Haven, Connecticut
  - Research Site, West Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Orlando, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Rosedale, Maryland
  - Research Site, Lincoln, Nebraska
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Gettysburg, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Germantown, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (14):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Créteil
  - Research Site, La Rochelle
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Jordan
  - Research Site, Kowloon
- Italy (6):
  - Research Site, Catania
  - Research Site, Cremona
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Ravenna
  - Research Site, Siena
- Poland (2):
  - Research Site, Gdynia
  - Research Site, Lodz
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Spain (7):
  - Research Site, A Coruña
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Valencia
- Taiwan (2):
  - Research Site, Chiayi City
  - Research Site, Taichung

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Aggarwal C, Martinez-Marti A, Majem M, Barlesi F, Carcereny E, Chu Q, Monnet I, Sanchez-Hernandez A, Dakhil S, Camidge DR, Pillet M, Brown M, Paliompeis C, Dowson A, Cooper ZA, Kumar R, Herbst RS. Durvalumab Alone or Combined With Novel Agents for Unresectable Stage III Non-Small Cell Lung Cancer: Update From the COAST Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2518440. doi: 10.1001/jamanetworkopen.2025.18440. PMID 40663352
- [Derived] Herbst RS, Majem M, Barlesi F, Carcereny E, Chu Q, Monnet I, Sanchez-Hernandez A, Dakhil S, Camidge DR, Winzer L, Soo-Hoo Y, Cooper ZA, Kumar R, Bothos J, Aggarwal C, Martinez-Marti A. COAST: An Open-Label, Phase II, Multidrug Platform Study of Durvalumab Alone or in Combination With Oleclumab or Monalizumab in Patients With Unresectable, Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Oct 10;40(29):3383-3393. doi: 10.1200/JCO.22.00227. Epub 2022 Apr 22. PMID 35452273
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9108C00001&attachmentIdentifier=de7dfeb7-8334-4784-8d4a-da8d429556aa&fileName=d9108c00001-csp-amendment-4_Redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9108C00001&attachmentIdentifier=51d2c3e5-8514-4a79-907b-da0a3149d00c&fileName=D9108C00001_Statistical_Analysis_Plan_v5_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9108C00001&attachmentIdentifier=f0bb70f9-6f4e-4554-b7e4-aafad3298d36&fileName=d9108c00001-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was randomized into the study on 3 January 2019 and the last participant was randomized on 6 July 2020.
Groups:
- Control Arm (Durvalumab Monotherapy): Durvalumab 1500 mg IV monotherapy Q4W
- Arm A (Durvalumab + Oleclumab): Durvalumab 1500 mg IV Q4W + Oleclumab 3000 mg IV (Q2W for cycles 1 and 2, then Q4W starting cycle 3)
- Arm B (Durvalumab + Monalizumab): Durvalumab 1500 mg IV Q4W + Monalizumab 750 mg IV Q2W
Period: Overall Study
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Started | 67 | 60 | 62
Completed | 21 | 29 | 30
Not Completed | 46 | 31 | 32
Not completed — Death | 27 | 23 | 24
Not completed — Lost to Follow-up | 6 | 2 | 1
Not completed — Withdrawal by Subject | 10 | 4 | 6
Not completed — Progressive Disease | 2 | 1 | 0
Not completed — Not Treated | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included participants who were randomized and were analyzed according to their randomized treatment group
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab) | Total
Number analyzed (Participants) | 67 | 60 | 62 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.9) | 63.8 (9.5) | 64.4 (9.2) | 64.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 20 | 60
  Male | 45 | 42 | 42 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 8
  Not Hispanic or Latino | 63 | 56 | 59 | 178
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 5 | 4 | 5 | 14
  Black or African American | 1 | 5 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 57 | 47 | 55 | 159
  Other | 1 | 2 | 0 | 3
  Missing | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: Participants]
  Canada | 3 | 2 | 1 | 6
  France | 15 | 19 | 5 | 39
  Hong-Kong | 1 | 2 | 3 | 6
  Italy | 0 | 3 | 3 | 6
  Portugal | 3 | 0 | 3 | 6
  Spain | 19 | 12 | 22 | 53
  Taiwan | 1 | 0 | 1 | 2
  United States | 25 | 22 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR) Rate as a Measure of Antitumor Activity of Durvalumab Alone vs Durvalumab in Combination With Novel Agents
Description: ORR was defined as the percentage of participants with at least one visit response of Complete Response (CR) or Partial Response (PR) per RECIST 1.1 for target lesions: CR: Disappearance of all target lesions; PR: >=30% decrease in the sum of the longest diameter of target lesions; OR = CR + PR.
Time Frame: ORR at 16 weeks after randomization is the timing for radiologic assessment of the primary endpoint
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 67 | 60 | 62
Percentage of Participants | 23.9 [14.3 to 35.9] | 35.0 [23.1 to 48.4] | 40.3 [28.1 to 53.6]

2. Secondary Outcome: Presence of Adverse Events as a Measure of Safety and Tolerability of Durvalumab Alone and in Combination With Novel Agents
Description: The secondary endpoint of safety as assessed by the presence of adverse events and serious adverse events
Time Frame: From time of signature of informed consent up to 15 months post the first dose of study treatment
Population: The As-treated population included all participants who receive any IP. Participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 66 | 59 | 61
Participants
  Participants with any TEAEs | 65 | 57 | 61
  Participants with any serious TEAEs | 23 | 20 | 17

3. Secondary Outcome: Presence of Clinically Significant Laboratory Values as a Measure of Safety and Tolerability of Durvalumab Alone and in Combination With Novel Agents
Description: The secondary endpoint of safety as assessed by the presence of Grade 3 or 4 clinical laboratory toxicities (based on NCI-CTCAE v5.0) in chemistry and hematology values
Time Frame: From baseline up to 15 months post the first dose of study treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 66 | 59 | 61
Participants
  Participants with any Grade 3 or 4 Alanine Aminostransferase (U/L) toxicities: number analyzed (Participants) | 64 | 56 | 60
  Participants with any Grade 3 or 4 Alanine Aminostransferase (U/L) toxicities | 1 | 0 | 0
  Participants with any Grade 3 or 4 Albumin (g/dL) toxicities: number analyzed (Participants) | 63 | 57 | 60
  Participants with any Grade 3 or 4 Albumin (g/dL) toxicities | 2 | 0 | 0
  Participants with any Grade 3 or 4 Amylase (U/L) toxicities: number analyzed (Participants) | 62 | 56 | 59
  Participants with any Grade 3 or 4 Amylase (U/L) toxicities | 1 | 0 | 2
  Participants with any Grade 3 or 4 Aspartate Aminotransferase (U/L) toxicities: number analyzed (Participants) | 64 | 57 | 60
  Participants with any Grade 3 or 4 Aspartate Aminotransferase (U/L) toxicities | 1 | 0 | 1
  Participants with any Grade 3 or 4 Creatinine (mg/dL) toxicities: number analyzed (Participants) | 64 | 57 | 60
  Participants with any Grade 3 or 4 Creatinine (mg/dL) toxicities | 1 | 0 | 0
  Participants with any Grade 3 or 4 Creatinine Clearance Rate (mL/min) toxicities: number analyzed (Participants) | 63 | 57 | 60
  Participants with any Grade 3 or 4 Creatinine Clearance Rate (mL/min) toxicities | 2 | 1 | 0
  Participants with any Grade 3 or 4 Gamma Glutamyl Transferase (U/L) toxicities: number analyzed (Participants) | 64 | 57 | 59
  Participants with any Grade 3 or 4 Gamma Glutamyl Transferase (U/L) toxicities | 1 | 0 | 0
  Participants with any Grade 3 or 4 Hyperkalemia (mEq/L) toxicities: number analyzed (Participants) | 64 | 57 | 60
  Participants with any Grade 3 or 4 Hyperkalemia (mEq/L) toxicities | 0 | 0 | 2
  Participants with any Grade 3 or 4 Hypokalemia (mEq/L) toxicities: number analyzed (Participants) | 64 | 57 | 60
  Participants with any Grade 3 or 4 Hypokalemia (mEq/L) toxicities | 1 | 0 | 1
  Participants with any Grade 3 or 4 Hypocalcemia (corrected) (mg/dL) toxicities: number analyzed (Participants) | 63 | 57 | 60
  Participants with any Grade 3 or 4 Hypocalcemia (corrected) (mg/dL) toxicities | 1 | 0 | 0
  Participants with any Grade 3 or 4 Hypernatremia (mEq/L) toxicities: number analyzed (Participants) | 64 | 57 | 60
  Participants with any Grade 3 or 4 Hypernatremia (mEq/L) toxicities | 1 | 2 | 1
  Participants with any Grade 3 or 4 Lipase (U/L) toxicities: number analyzed (Participants) | 63 | 56 | 60
  Participants with any Grade 3 or 4 Lipase (U/L) toxicities | 1 | 4 | 2
  Participants with any Grade 3 or 4 Hemoglobin increased (g/dL) toxicities: number analyzed (Participants) | 64 | 57 | 58
  Participants with any Grade 3 or 4 Hemoglobin increased (g/dL) toxicities | 3 | 0 | 0
  Participants with any Grade 3 or 4 Lymphocyte count increased (10^3/uL) toxicities: number analyzed (Participants) | 64 | 57 | 58
  Participants with any Grade 3 or 4 Lymphocyte count increased (10^3/uL) toxicities | 19 | 11 | 11
  Participants with any Grade 3 or 4 Platelet count decreased (10^3/uL) toxicities: number analyzed (Participants) | 64 | 57 | 58
  Participants with any Grade 3 or 4 Platelet count decreased (10^3/uL) toxicities | 1 | 0 | 0

4. Secondary Outcome: Presence of Abnormalities in Vital Signs as a Measure of Safety and Tolerability of Durvalumab Alone and in Combination With Novel Agents
Description: The secondary endpoint of safety as assessed by the presence of abnormal vital signs reported as adverse events
Time Frame: From baseline up to 15 months post the first dose of study treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 66 | 59 | 61
Participants
  Hypertension | 3 | 3 | 0
  Hypotension | 2 | 0 | 3
  Palpitations | 0 | 0 | 1
  Pyrexia | 6 | 8 | 10
  Tachycardia | 1 | 2 | 2

5. Secondary Outcome: Duration of Response (DoR) as a Measure of Efficacy of Durvalumab Alone vs Durvalumab in Combination With Novel Agents
Description: The duration from the first documentation of a subsequently confirmed OR to the first documentation of a disease progression according to RECIST v1.1 or death due to any cause, whichever occurs first. Only participants who have achieved OR (confirmed CR or confirmed PR) will be evaluated for DoR
Time Frame: Up to approximately 54 months (through the database cutoff date of 18-Jul-2023).
Population: The Intent-to-treat (ITT) population included participants who were randomized and were analyzed according to their randomized treatment group. Only participants with an objective response were included in the DoR analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 16 | 21 | 25
Months | NA [14.1 to NA] — The median and upper limit of 95% CI could not be calculated as they were not reached. | 29.9 [17.1 to NA] — The upper limit of 95% CI could not be calculated as it was not reached. | 23.0 [10.2 to NA] — The upper limit of 95% CI could not be calculated as it was not reached.

6. Secondary Outcome: Disease Control (DC) as a Measure of Efficacy of Durvalumab Alone vs Durvalumab in Combination With Novel Agents
Description: Disease control rate (DCR) was defined as the percentage of participants with a BOR of confirmed CR, confirmed PR, or SD (maintained for ≥ 16 weeks) based on RECIST v1.1.
Time Frame: Up to approximately 54 months (through the database cutoff date of 18-Jul-2023).
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 67 | 60 | 62
Percentage of Participants | 58.2 [45.5 to 70.2] | 80.0 [67.7 to 89.2] | 79.0 [66.8 to 88.3]

7. Secondary Outcome: Progression-Free Survival (PFS) as a Measure of Efficacy of Durvalumab Alone vs Durvalumab in Combination With Novel Agents
Description: PFS was defined as the time from randomization until the first documentation of disease progression according to RECIST v1.1 or death due to any cause, whichever occurs first
Time Frame: Up to approximately 54 months (through the database cutoff date of 18-Jul-2023).
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 67 | 60 | 62
Months | 7.3 [4.0 to 13.8] | 21.1 [10.4 to 30.9] | 19.8 [13.6 to 31.3]

8. Secondary Outcome: Progression-Free Survival 12 Month Landmark Rate (PFS-12) as a Measure of Efficacy of Durvalumab Alone vs Durvalumab in Combination With Novel Agents
Description: PFS-12 was defined as the percentage of participants who were alive and progression free at 12 months after randomization.
Time Frame: PFS rate at 12 months after randomization.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 67 | 60 | 62
Percentage of Participants | 37.6 [24.7 to 50.4] | 63.5 [49.2 to 74.7] | 73.2 [59.6 to 82.9]

9. Secondary Outcome: Overall Survival (OS) as a Measure of Efficacy of Durvalumab Alone vs Durvalumab in Combination With Novel Agents
Description: OS was defined as the time from the date of randomization until death due to any cause.
Time Frame: From time of randomization until death due to any cause. Assessed through the database cutoff date of 18-Jul-2023).
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 67 | 60 | 62
Months | 40.9 [22.6 to NA] — The upper limit of 95% CI could not be calculated as it was not reached. | NA [31.9 to NA] — The median and upper limit of 95% CI could not be calculated as they were not reached. | NA [31.3 to NA] — The median and upper limit of 95% CI could not be calculated as they were not reached.

10. Secondary Outcome: Pharmacokinetics of Durvalumab Alone and in Combination With Novel Agents
Description: Geometric mean serum concentrations of durvalumab (μg/mL) were reported for each time point where data warrant, as appropriate.
Time Frame: From randomization up to 15 months after first treatment: Cycle 1 Day 1 pre-dose and at end of infusion, Cycle 2 Day 1 pre-dose (1 month), Cycle 7 Day 1 pre-dose (6 months), Cycle 11 Day 1 pre-dose (10 months) and 15 months post Cycle 1 Day 1
Population: The PK-evaluable durvalumab population included participants from the As-treated population who had a non-missing baseline PK durvalumab concentration and at least one non-missing post-baseline PK durvalumab concentration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 57 | 41 | 51
Micrograms per milliliter
  Cycle 1 Day 1: End of Infusion: number analyzed (Participants) | 52 | 34 | 46
  Cycle 1 Day 1: End of Infusion | 318.0 (199.6) | 277.4 (316.1) | 223.7 (1272)
  Cycle 2 Day 1: Pre-Dose: number analyzed (Participants) | 48 | 37 | 47
  Cycle 2 Day 1: Pre-Dose | 59.7 (58.6) | 68.0 (49.9) | 74.3 (40.7)
  Cycle 7 Day 1: Pre-Dose: number analyzed (Participants) | 25 | 29 | 35
  Cycle 7 Day 1: Pre-Dose | 151.6 (37.7) | 127.9 (66.4) | 176.5 (45.6)
  Cycle 11 Day 1: Pre-Dose: number analyzed (Participants) | 16 | 22 | 31
  Cycle 11 Day 1: Pre-Dose | 156.7 (50.0) | 146.5 (91.3) | 172.4 (40.4)

11. Secondary Outcome: Pharmacokinetics of Novel Agents in Combination With Durvalumab
Description: Geometric mean serum concentrations of oleclumab (μg/mL) and monalizumab (μg/mL) were reported for each time point where data warrant, as appropriate.
Time Frame: as for outcome 10
Population: The PK-evaluable oleclumab/monalizumab population included participants from the As-treated population who had a non-missing baseline PK oleclumab/monalizumab concentration and at least one non-missing post-baseline PK oleclumab/monalizumab concentration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 52 | 51
Micrograms per milliliter
  Cycle 1 Day 1: End of Infusion: number analyzed (Participants) | 52 | 49
  Cycle 1 Day 1: End of Infusion | 581.6 (210.5) | 160.0 (286.4)
  Cycle 2 Day 1: Pre-Dose: number analyzed (Participants) | 37 | 43
  Cycle 2 Day 1: Pre-Dose | 216.4 (58.6) | 102.6 (39.2)
  Cycle 7 Day 1: Pre-Dose: number analyzed (Participants) | 37 | 32
  Cycle 7 Day 1: Pre-Dose | 124.5 (109.0) | 194.5 (33.8)
  Cycle 11 Day 1: Pre-Dose: number analyzed (Participants) | 26 | 30
  Cycle 11 Day 1: Pre-Dose | 132.0 (166.8) | 196.2 (48.7)

12. Secondary Outcome: Presence of Detectable Anti-Drug Antibody (ADA) Response to Durvalumab Alone and in Combination With Novel Agents
Description: ADA prevalence was defined as the percentage of participants with positive ADA result at any time, baseline or post-baseline. ADA positive post-baseline only was also referred to as treatment-induced ADA positive. Treatment-boosted ADA was defined as baseline positive ADA titer that was boosted to a 4-fold or higher following drug administration. Persistently positive was defined as positive at ≥2 post-baseline assessments (with ≥16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive.
  ADA incidence (treatment-emergent ADA positive) was defined as the sum of treatment-induced ADA and treatment-boosted ADA.
Time Frame: From randomization up to 15 months after first treatment: Cycle 1 Day 1 pre-dose, Cycle 2 Day 1 pre-dose (1 month), Cycle 7 Day 1 pre-dose (6 months), Cycle 11 Day 1 pre-dose (10 months) and 15 months post Cycle 1 Day 1
Population: The durvalumab ADA-evaluable population included participants from the As-treated population who had a non-missing baseline durvalumab ADA result and at least one non-missing post-baseline durvalumab ADA result
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm (Durvalumab Monotherapy) | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 40 | 18 | 33
Participants
  ADA positive at any visit (ADA prevalence) | 3 | 1 | 2
  Treatment-emergent ADA positive (ADA incidence) | 1 | 0 | 0
  Treatment-boosted ADA | 0 | 0 | 0
  Treatment-induced ADA (positive post-baseline only) | 1 | 0 | 0
  ADA positive at baseline only | 2 | 1 | 2
  ADA positive post-baseline and positive at baseline | 0 | 0 | 0
  Persistently positive | 1 | 0 | 0
  Transiently positive | 0 | 0 | 0

13. Secondary Outcome: Presence of Detectable Anti-Drug Antibody (ADA) Response to Novel Agents in Combination With Durvalumab
Description: as for outcome 12
Time Frame: as for outcome 12
Population: The oleclumab/monalizumab ADA-evaluable population included participants from the As-treated population who had a non-missing baseline oleclumab/monalizumab ADA result and at least one non-missing post-baseline oleclumab/monalizumab ADA result
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Durvalumab + Oleclumab) | Arm B (Durvalumab + Monalizumab)
Number analyzed (Participants) | 54 | 51
Participants
  ADA positive at any visit (ADA prevalence) | 0 | 1
  Treatment-emergent ADA positive (ADA incidence) | 0 | 1
  Treatment-boosted ADA | 0 | 0
  Treatment-induced ADA (positive post-baseline only) | 0 | 1
  ADA positive at baseline only | 0 | 0
  ADA positive post-baseline and positive at baseline | 0 | 0
  Persistently positive | 0 | 0
  Transiently positive | 0 | 1

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from time of signature of informed consent up to 15 months post the first dose of study treatment
Description: Treatment-emergent adverse events (TEAEs) are defined as events present at baseline that worsen in intensity after administration of study IP or events absent at baseline that emerge after administration of study IP. All TEAEs that occurred on and after first dose up to 3 months after last dose of IP (any) were summarized.
Groups:
- Durvalumab Monotherapy; Durvalumab + Oleclumab; Durvalumab + Monalizumab: Description (Arm-group)
Arm/Group | Durvalumab Monotherapy | Durvalumab + Oleclumab | Durvalumab + Monalizumab
All-Cause Mortality (participants affected / at risk) | 27/66 | 23/59 | 24/61
Serious Adverse Events (participants affected / at risk) | 23/66 | 20/59 | 17/61
Other Adverse Events (participants affected / at risk) | 61/66 | 52/59 | 58/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Monotherapy (N=66) | Durvalumab + Oleclumab (N=59) | Durvalumab + Monalizumab (N=61)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Monotherapy (N=66) | Durvalumab + Oleclumab (N=59) | Durvalumab + Monalizumab (N=61)
Hypertension (Vascular disorders) | 3 (4) | 3 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 10 (11) | 8 (8) | 13 (14)
Dry eye (Eye disorders) | 1 (1) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (10) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 8 (8) | 13 (19)
Nausea (Gastrointestinal disorders) | 8 (10) | 1 (1) | 5 (7)
Anaemia (Blood and lymphatic system disorders) | 5 (8) | 5 (9) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 3 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (5) | 5 (6) | 5 (5)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 6 (8) | 7 (8) | 9 (10)
Bronchitis (Infections and infestations) | 1 (1) | 4 (9) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 4 (4) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 6 (8) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (7) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 5 (6)
Headache (Nervous system disorders) | 2 (2) | 4 (5) | 5 (5)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 19 (22) | 26 (29)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (7) | 8 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (9) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 10 (17) | 15 (18)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 9 (14) | 8 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 5 (5)
Hyperthyroidism (Endocrine disorders) | 9 (10) | 7 (7) | 6 (6)
Pneumonia (Infections and infestations) | 5 (7) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (7) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (3) | 4 (7)
Amylase increased (Investigations) | 7 (13) | 4 (5) | 5 (7)
Lipase increased (Investigations) | 6 (11) | 5 (6) | 5 (5)
Lymphocyte count decreased (Investigations) | 4 (7) | 8 (14) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 6 (6) | 5 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (15) | 10 (10) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (7) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 6 (6)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (4) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 15 (20) | 14 (18)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (5)
Asthenia (General disorders) | 10 (11) | 11 (12) | 15 (16)
Fatigue (General disorders) | 7 (8) | 7 (8) | 9 (9)
Blood creatinine increased (Investigations) | 4 (5) | 0 (0) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT03822351/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT03822351/SAP_003.pdf